CLINICAL TRIAL: NCT03211104
Title: Comparison of Duration of Treatment Interruption With or Without Curcumin During the Off Treatment Periods in Patients With Prostate Cancer Undergoing Intermittent Androgen Deprivation Therapy : a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Comparison of Duration of Treatment Interruption With or Without Curcumin During the Off Treatment Periods in Patients With Prostate Cancer Undergoing Intermittent Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-06-068
Record Dates: First submitted 2017-05-09; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: intermittent androgen deprivation therapy; curcumin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- curcumin (Experimental): Curcumin extracted from curcuma longa linn.
  * formulation : curcumin powder 240mg/capsule
  * general name : Diferuloylmethane
  Taking curcumin 3 times a day(1,440mg/day) for 6 months at the first off treatment in patients with prostate cancer receiving intermittent androgen deprivation therapy
  Interventions: Dietary Supplement: curcumin
- control (Placebo Comparator): The control group Take a placebo containing lactose and vitamin B2. Reddish brown capsules with the same shape as curcumin.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: curcumin
  Arms: curcumin
Dietary Supplement: Placebo
  Arms: control

SUMMARY:
This was a placebo-controlled, double-blind, randomized trial designed with the aim of establishing whether curcumin influenced the duration of treatment interruption and rate of prostatic specific antigen(PSA) progression, compared with placebo among men with prostate cancer receiving intermittent androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with prostate cancer in biopsy
* among patients with biochemical recurrence after treatment(radical prostatectomy, radiation therapy, focal therapy, etc.) for localized prostate cancer or metastatic prostate cancer at the time of diagnosis, who received intermittent androgen deprivation therapy(IAD)
* patients who off-treatment for the first time by receiving androgen deprivation therapy(ADT) for more than 6 months and PSA nadir remained stable for more than 3 months

Exclusion Criteria:

* previous history of IAD
* patient with other serious or ongoing medical or psychiatric disease other than prostate cancer
* hypersensitivity or suspicious of curcumin
* history of taking health supplements containing curcumin for prostate cancer treatment before 6 months of clinical trial participation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-08-30 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2015-08-05 (Actual)

PRIMARY OUTCOMES:
Duration of treatment interruption with or without curcumin | up to 42 months
  To determine whether the period from the first interruption of the androgen deprivation therapy to the time when androgen deprivation therapy needs to be retreated differ between curcumin group and placebo group

SECONDARY OUTCOMES:
Mean change in PSA(ng/ml) from baseline between curcumin group versus placebo | 0,1,2,3,4,5,6,12,18,30,42 months
  Measure the mean change of PSA at each point from the baseline and compare differences between the two groups
Mean change in testosterone(ng/ml) from baseline between curcumin group versus | 0,1,2,3,4,5,6,12,18,30,42 months
  Measure the mean change of testosterone at each point from the baseline and compare differences between the two groups
Adverse events | 0,1,2,3,4,5,6,12,18,30,42 months
  Adverse events were recorded according to the Common Terminology Criteria for Adverse Events(CTCAE). Vital sign, blood test and urine analysis were also performed.

REFERENCES:
- [Background] Cloughesy T, Finocchiaro G, Belda-Iniesta C, Recht L, Brandes AA, Pineda E, Mikkelsen T, Chinot OL, Balana C, Macdonald DR, Westphal M, Hopkins K, Weller M, Bais C, Sandmann T, Bruey JM, Koeppen H, Liu B, Verret W, Phan SC, Shames DS. Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase II Study of Onartuzumab Plus Bevacizumab Versus Placebo Plus Bevacizumab in Patients With Recurrent Glioblastoma: Efficacy, Safety, and Hepatocyte Growth Factor and O6-Methylguanine-DNA Methyltransferase Biomarker Analyses. J Clin Oncol. 2017 Jan 20;35(3):343-351. doi: 10.1200/JCO.2015.64.7685. Epub 2016 Dec 5. PMID 27918718
- [Background] van Die MD, Bone KM, Emery J, Williams SG, Pirotta MV, Paller CJ. Phytotherapeutic interventions in the management of biochemically recurrent prostate cancer: a systematic review of randomised trials. BJU Int. 2016 Apr;117 Suppl 4(Suppl 4):17-34. doi: 10.1111/bju.13361. Epub 2016 Feb 22. PMID 26898239